

#### PM104-B-001-09

Phase II Clinical and Pharmacokinetic Trial of Zalypsis® in Patients with Advanced and/or Metastatic Endometrial or Cervical Cancer Treated with at least One Line of Systemic Therapy

# **Statistical Analysis Plan**

Author Mariano Siguero, Biostatistician

Version 1.0

**Date** 28-07-09 **NCT Code** 00900562

# **Table of contents**

| 1 | INT | TRODUCTION5 |
|---|-----|---------------------------------------------------------------|
| | 1.1 | Study rationale5 |
| | 1.2 | Information on Study Drug5 |
| 2 | OB. | JECTIVES5 |
| | 2.1 | Primary5 |
| | 2.2 | Secondary5 |
| 3 | STU | JDY DESIGN5 |
| 4 | STU | JDY POPULATIONS6 |
| | 4.1 | Analysis populations |
| | | Afficacy population 6 afety population 6 |
| 5 | ENI | DPOINTS6 |
| | 5.1 | Primary endpoints6 |
| | 5.2 | Secondary endpoints |
| 6 | SAN | MPLE SIZE7 |
| | 6.1 | Sample size determination |
| | 6.2 | Interim analyses |
| 7 | STA | ATISTICAL ANALYSIS9 |
| | 7.1 | Treatment discontinuation and protocol deviations management9 |
| | 7.2 | Demographic analysis9 |
| | 7.3 | Exposure |
| | 7.4 | Statistical methodology for efficacy |
| | 7.5 | Statistical methodology for safety10 |
| | 7.6 | Missing values management11 |
| 8 | PH | ARMACOKINETIC (PK) AND PHARMACOGENOMIC (PGX) EVALUATION11 |

| 9 | S | TATISTICAL SOFTWARE | 11 |
|---|---|---|---|
| 10 | A | PPENDIX I. PATIENTS DISPOSITION | 12 |
| | 10.1 | General characteristics | 12 |
| | 10.1.1 | Patients treated, eligible and evaluable | 12 |
| | | Reasons for treatment discontinuation. | |
| | | Protocol deviations | |
| 11 | A | PPENDIX II. EFFICACY EVALUATION | 14 |
| | 11.1 | Baseline characteristics | 14 |
| | 11.1.1 | Patients characteristics at baseline | 14 |
| | | Histology and time from diagnosis | |
| | | Prior anticancer therapy | |
| | | Prior history | |
| | | Physical examination, vital signs, electrocardiogram and other tests | |
| | | Hematological values at baseline | |
| | | Biochemical values at baseline | |
| | | Other metabolic values at baseline | |
| | | Signs and symptoms at baseline | |
| | | Concomitant therapy | |
| | 11.2.2<br>11.2.3 | Response | 21<br>23<br>24 |
| 12 | A.<br>12.1 | PPENDIX III. SAFETY EVALUATION Extent of exposure | |
| | 12 1 1 | Treatment administration | 24 |
| | | Dose delays | |
| | | • | |
| | | Dose reduction | |
| | 12.2 | Toxicity | 28 |
| | 12.2.1 | Adverse events | 28 |
| | | Serious toxicity rate | |
| | | Serious adverse events | |
| | 12.3 | Laboratory evaluation | 29 |
| | 12.3.1 | Hematological abnormalities | 29 |
| | | Biochemistry abnormalities | |
| | | Other metabolic abnormalities | |

| | 12.4 | Vital Signs |
|----|------|-----------------------------------------|
| | 12.5 | Concomitant medication during treatment |
| 13 | FIG | SURES |

#### 1 Introduction

## 1.1 Study rationale

This Statistical Analysis Plan (SAP) explains in detail the statistical analyses that will be carried out for Pharmamar in PM104 - B - 001 - 09 study. The analyses described in this SAP are based upon and supplement those described in the study protocol (dated 27-Jan-2009).

## 1.2 Information on Study Drug

PM00104 is a new synthetic alkaloid that has been selected for clinical development based on its in vitro activity against human solid and non-solid tumor cell lines, its in vivo activity in xenografted human tumors, as well as an acceptable non-clinical toxicology profile.

# 2 Objectives

The study protocol states the following:

## 2.1 Primary

• To evaluate the antitumor activity of PM00104 administered as a 1-hour intravenous (i.v) infusion on Day 1, 8 and 15 every four weeks (d1, d8 and d15; q4wk) to patients with advanced and/or metastatic endometrial or cervical cancer previously treated with one line of systemic chemotherapy.

#### 2.2 Secondary

- To determine the safety profile of this PM00104 regimen in these patients.
- To determine the pharmacokinetic (PK) profile of this PM00104 regimen in these patients.
- To determine the pharmacogenomic (PGx) profile of this PM00104 regimen in these patients. Hypothesis-generating exploratory PGx analyses will be conducted to correlate the molecular parameters found in the tumor samples of the patients with the clinical results achieved with PM00104

## 3 Study design

Multicenter, open label, phase II clinical trial with single-agent PM00104 given as a as a 1-hour i.v. infusion on d1, d8 and d15 q4wk to patients with advanced and/or metastatic endometrial or cervical cancer progressing after at least one line of systemic chemotherapy.

The primary endpoint of the study is the overall response rate (ORR), defined as the percentage of patients with objective response (OR; complete or partial response) as defined by the Response Evaluation Criteria in Solid Tumors (RECIST).

#### 4 Study populations

## 4.1 Analysis populations

Female adult patients with endometrial (Group 1) or cervical cancer (Group 2) progressing after at least one previous line of systemic chemotherapy are eligible for this trial. To be included in the study, patients have to fulfill all inclusion criteria and none of the exclusion criteria.

#### 4.1.1 Efficacy population

To be evaluable for efficacy, patients must have received at least four infusions of the six infusions in the first two cycles and at least one disease measurement recorded not less than six weeks after treatment onset will be evaluable for efficacy.

In addition, any eligible patient who receives at least two of the three infusions in one treatment cycle and experience disease progression or die due to progressive disease (PD) prior to response evaluation will be considered evaluable for the main endpoint (ORR) and will be categorized as an "early progression".

Patients withdrawn due to toxicity without any tumor assessment after the start of study treatment will be considered as "treatment failures" and will not be replaced.

Patients withdrawn due to significant clinical deterioration of unknown reason, hypersensitivity reactions, refusal to continue on study for any reason or unrelated AEs without any tumor assessment after the start of study treatment will be considered not evaluable for efficacy and will be replaced.

## 4.1.2 Safety population

All patients who have received at least one complete or partial infusion of PM00104 infusion will be included in the safety analysis.

#### 5 Endpoints

## 5.1 Primary endpoints

Overall response rate (ORR), defined as the percentage of patients with confirmed objective response (OR), either complete (CR) or partial (PR) response according to the RECIST.

## 5.2 Secondary endpoints

- Progression-free survival at four months (PFS4 rate), defined as the percentage of patients who
  are alive and with no evidence of disease progression at four months after the first study drug
  administration.
- Progression-free survival rate at six months (PFS6), defined as the percentage of patients who are alive and with no evidence of disease progression at six months after the first study drug administration.
- Duration of response (DR), defined as the time between the date when the response criteria (PR or CR, the first that is reached) are fulfilled and the first date when disease progression, recurrence or death is objectively documented (taking the smallest measurements documented since the treatment started as reference for progressive disease).

- Progression-free survival (PFS), defined as the time from the first day of study treatment to the day of negative assessment (progression or death) or last tumour evaluation.
- Overall survival (OS), defined as the time from the first day of treatment to the date of death (or the last day when the patient is known to be alive). Survival will be followed for up to six months after the treatment discontinuation of the last patient.
- Safety profile: AEs, SAEs, laboratory evaluations, deaths and the reason for study discontinuations, dose delays, modifications or omissions will be analyzed. All AEs and SAEs will be classified according to the NCI-CTCAE, version 3.0, and will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 10.0.

#### • Treatment exposure:

- Date of treatment start: Date of treatment dose at cycle 1.
- Date of last dose: Date of last treatment dose at last cycle.
- Date of treatment discontinuation (for the purpose of exposure calculations): The minimum date between the death date and the date of the first infusion of last cycle + 28 days.
- Body Surface Area (BSA): The calculated surface of a human body measured in m<sup>2</sup>.
- *Treatment duration*: The time between the day of the first dose and the day of treatment discontinuation (in weeks).
- *Total cumulative dose*: The sum of all the PM00104 doses from the first cycle until last cycle including the dose received in last cycle. (Expressed in mg/m²).
- *Absolute dose intensity:* The actual cumulative dose divided by number of weeks of treatment. (Expressed in mg/m²/wk).
- *Intended dose intensity*: The planned dose per cycle divided by the planned weeks by cycle. (Expressed in mg/m²/wk).
- Relative dose intensity: The ratio of absolute dose intensity (x100) divided by the intended dose intensity. (Expressed in percentage).
- Pharmacokinetic/Pharmacodynamic parameters.
- Pharmacogenomic profile

# 6 Sample size

#### 6.1 Sample size determination

In this phase II trial, efficacy of PM00104 will be evaluated in two different groups of patients with endometrial or cervical cancer.

Group 1 (endometrial cancer): A Simon two-stage design will be adopted in this group to test the null hypothesis that the ORR by RECIST is  $\leq 10\%$  versus the alternative that ORR  $\geq 30\%$  (two-sided test; alpha=0.1 and beta=0.1).

A maximum of 30 evaluable patients will be included in this group. In a first stage, 10 evaluable patients will be recruited. If one or more  $(\geq 1)$  patients achieve an objective response, the accrual in this group will be expanded with 20 additional evaluable patients.

If the total number of patients with objective response is 6 or more ( $\geq$  6) in 30 evaluable patients (i.e., an ORR in the whole study of at least 20%), the null hypothesis will be rejected and PM00104 will be considered for further clinical development in endometrial cancer.

Group 2 (cervical cancer): Also a Simon two-stage design where the null hypothesis ORR by RECIST is  $\leq 5\%$  vs. ORR  $\geq 20\%$  (two-sided test; alpha=0.1 and beta=0.1).

A maximum of 32 evaluable patients will be included in this group. In a first stage, 18 evaluable patients will be recruited. If one or more ( $\geq 1$ ) patients achieve an objective response, the accrual in this group will be expanded with 14 additional evaluable patients.

If the total number of patients with objective response is 4 or more ( $\geq$  4) in 32 evaluable patients (i.e., an ORR in the whole study of at least 12.5%), the null hypothesis will be rejected and PM00104 will be considered for further clinical development in cervical cancer.

#### 6.2 Interim analyses

Interim efficacy analysis will be performed when the 10 first evaluable patients have been recruited in the group 1 and 18 patients have been recruited in the group 2. In addition, a safety evaluation will be performed when 10 patients in each group will be recruited and followed for at least four weeks. The study will be stopped, and the recommended dose re-evaluated if the stopping rule described below is met in any of the groups.

Other non-scheduled interim analyses might be performed exclusively for enhancing the safety of the patients.

Early stopping rule:

An early stopping rule for excessive toxicity will be evaluated when ten patients in each group will be recruited and followed for at least four weeks. A "serious toxicity" rate (STR) of 40% or more will be considered inadequate. The following are considered serious toxicities:

- Drug-related grade 4 neutropenia lasting for more than seven days.
- Grade 4 thrombocytopenia.
- Grade 3/4 nausea/vomiting despite adequate prophylaxis.
- Grade 3/4 transaminase increase lasting for more than seven days.
- Grade 3/4 fatigue.
- Any other grade 3/4 drug-related event leading to early study discontinuation.

If  $\geq$  4 patients of the first 10 patients had one of these serious toxicities, the trial will be stopped and the recommended dose and/or administration schedule for phase II will be re-evaluated. With this stopping rule, the probability of  $\geq$ 4/10 STR in the sample (if the true probability of STR is <1/6) is 0.0697. On the other hand, the probability of observing  $\leq$ 3/10 STR in the sample (if the true probability of STR is >40%) would be 0.3822.

#### 7 Statistical analysis

## 7.1 Treatment discontinuation and protocol deviations management

The accrual and study discontinuation details will be presented descriptively. The reasons for treatment discontinuation will be described by counts and percentages, overall and by number of cycles received. Reasons of treatment discontinuation other than disease progression will be detailed.

A study of the protocol deviations deemed relevant according to the Data Management Plan and Oncology review will be made following the ICH guidelines. The protocol deviations will be listed by type of deviation:

- Patients entered but not satisfying entry criteria
- Patients developing withdrawal criteria but not withdrawn
- Patients receiving incorrect dose or schedule
- Patients receiving excluded concomitant treatment

## 7.2 Demographic analysis

Demographics and baseline characteristics will be summarized by group for all recruited patients.

Continuous variables will be summarized and presented with summary statistics, i.e., median and range, mean, standard deviation,.

Categorical variables will be summarized in frequency tables. Percentages in the summary tables will be rounded and may therefore not always add up to exactly 100%.

In case of pre-treatment characteristics with multiple measurements per patient before the start of treatment (laboratory assessments, vital signs) the baseline measurement will be considered the last value prior to or on the first day of treatment.

Age, sex, race, baseline weight, height, body surface area (BSA), PS, pulse, BPS, BPD, temperature, LVEF, ECG and X-ray results will be summarized descriptively. Age is calculated based on the date of birth at the time date of registration date.

For solid tumors, histology diagnosis, number of organs involved and sites of disease will be described following standard tables detailed in section 10 (Appendix I).

A frequency tabulation of the number of patients with the different types of previous cancer surgery, radiotherapy and systemic therapy will be given.

A summary of prior relevant history and signs and symptoms will be presented per patient.

Laboratory values at baseline will be tabulated. Median values, ranges and CTC grades will be displayed by laboratory parameters.

Concomitant therapies will be categorized per ATC (level 1 and 4) class and coded term. The number of patients receiving each type of therapy during the treatment phase will be tabulated in 2 separate tables: a frequency tabulation of the different therapies that started pre-study, and a frequency tabulation of the different therapies that started during the study. Each table will be

generated once by class, and once by coded term. The accompanying listing will contain all concomitant therapies.

## 7.3 Exposure

Cumulative dose, dose intensity and relative dose intensity, cycle delay, and dose modifications or omissions will be described following standard tables detailed in section 12 (Appendix III).

#### 7.4 Statistical methodology for efficacy

Binomial estimates with exact 95% CIs will be calculated for the analysis of the main endpoint (ORR) and the secondary endpoints PFS4 and PFS6 rates. Time-to-event endpoints (DR, PFS and OS) will be analyzed according to the Kaplan-Meier method.

If relevant, efficacy parameters versus baseline covariates will be analyzed and appropriate test will be used (i.e., the Fisher exact test for categorical variables, the log-rank test or Cox regression for time-to-event variables, etc.).

The characteristics of patients with complete response, partial response, or free from progression at 4 months, will be described.

Statistical tests, if and when they are carried out, will only have an exploratory purpose and have a threshold of  $\alpha = 5\%$ . Exact binomial Confidence Intervals will be calculated with the same significance level.

See section 11 (Appendix II) for further details on the efficacy analysis.

#### 7.5 Statistical methodology for safety

Descriptive statistics, tabulation and graphic representation will be used for the evaluation of safety by tumor type in this phase II study, as described in section 12 (Appendix III).

If the safety profile of PM00104 is similar in both study groups (endometrial and cervical cancer), a pooled analysis for all included patients regardless its tumor type could be performed for safety.

Adverse events will be graded according to NCI-CTCAE version 3.0. The incidence and grade of adverse events and laboratory abnormalities will be calculated considering the most severe grade per patient and cycle.

Descriptive statistics will be used to present the profiles of drug-related adverse events, drug-related deaths, SAE and drug-related treatment discontinuation and the observed grade 1-4 toxicities, per patient and per cycle.

The shift of severity grades from baseline to the worst occurrence during treatment will be tabulated. The time to onset and recovery from neutrophils, platelets and hepatic enzymes elevations will be illustrated by means of descriptive statistics.

Database listings of deaths and serious adverse events will be provided, including at least date of onset and resolution (if applicable), severity, relationship to study drug, significant consequences and actions taken.

PS, weight gain – loss and LVEF measurements evolution during the study will be summarized by frequency tabulation.

See section 12 (Appendix III) for further details on the safety analysis.

#### 7.6 Missing values management

In case of missing values in the determination of protocol deviations (i.e. time from last anticancer treatment to start of treatment with PM00104) the most conservative approach will be taken for the evaluation.

If a date is missing, the worst case will be taken into account when calculating the difference between two dates. In such a case, this will be specified in the table footnote.

The cycles with missing information regarding laboratory values or adverse events will be subtracted from the denominator of the tables.

As regards of the analysis of Time to Progression, in case of more than one missing tumor scan between the last evaluation without progression and the documentation of progressive disease, the time to progression will be censored at the day of the last tumor evaluation without progression.

## 8 Pharmacokinetic (PK) and pharmacogenomic (PGx) evaluation

These analysis will be described in two different documents not included in this SAP.

#### 9 Statistical software

Oracle Clinical will be used for double data entry and clinical data management.

SAS v8.2 will be used for all the statistical analysis.

## TABLES, LISTINGS AND FIGURE SHELLS

**NOTE:** All tables, listings and figures described in this section will be duplicated in two different groups. First, patients with endometrial cancer (group 1) and secondly, patients with cervical cancer (group 2).

If appropriate, a pooled analysis for all included patients regardless its tumor type (group 1 + group 2) could be performed for Safety as in Sections 12.2 and 12.3.

Each particular table, listing and figure will have a comprehensive header and/or footnotes, identifying the group of treatment and/or relevant specifications.

## 10 Appendix I. Patients disposition.

#### 10.1 General characteristics.

#### 10.1.1 Patients treated, eligible and evaluable.

Table 10.1.1. 1. Patients accrual by institution.

| | Inc | titution 1 | Inst | itution 2 | Institu | ution | 7 | otal |
|---|---|---|---|---|---|---|---|---|
| | 1115 | utuuon 1 | 11151 | itution 2 | 1115111 | uuon | 1 | otai |
| | N | % | N | % | N | % | N | % |
| N-included | | | | | | | | |
| N-treated | | | | | | | | |

Table 10.1.1. 2. Disposition of patients.

| Event | Date |
|----------------------------------|------|
| Date first consent | |
| Date first dose of first patient | |
| Date last consent | |
| Date first dose of last patient | |
| Date last dose | |
| Last follow up date | |

Table 10.1.1. 3. Number of patients evaluable for analysis.

| _ | | valuable<br>efficacy | N.evaluable<br>for safety | | Total | |
|---|---|---|---|---|---|---|
| | $\mathbf{N}$ | % | N | % | $\mathbf{N}$ | % |
| N-included | | | | | | |
| N-treated | | | | | | |

## 10.1.2 Reasons for treatment discontinuation.

Table 10.1.2. 1. Reasons for treatment discontinuation.

| Progressive disease | | | | | | | MT91 | |
|---|---|---|---|---|---|---|---|---|
| Progressive disease | | | | | | N | tal | % |
| | | | | | | = ' | | , • |
| Patient refusal | | | | | | | | |
| Investigator decision | | | | | | | | |
| Other* | | | | | | | | |
| See Listing 10.1.2.5 | | | | | | | | |
| .hl. 10 1 2 2 D | 4 4 . 4 | 4: 4 | : <b>1</b> | l £1 | | 1 | | |
| able 10.1.2. 2. Reasons for tre | aument un | scommuai | ion by nu | Last Cycl | | | | |
| | | ycle 1 | <u> </u> | ycle 2 | | cle (X) | | Total |
| | $\frac{\mathcal{L}}{N}$ | <u>%</u> | N | <del>yeie 2</del><br>% | N | % | N | % |
| Progressive disease | 11 | , 0 | 11 | , 0 | 11 | 7.0 | - ' | , 0 |
| Patient refusal | | | | | | | | |
| Investigator decision | | | | | | | | |
| Other* | | | | | | | | |
| See Listing 10.1.2.5 | | | | | | | | |
| able 10.1.2. 3 Reason for end | of study. | | | | | | | |
| | | | | | | <u>T</u> | otal | % |
| Toxicity (study drug) Death Other See Listing 10.1.2.6 | | | | | | | | |
| able 10.1.2. 4. Time on treatm | | | | | | | | |
| | | <u>N</u> | M | ledian | | Min | | Max |
| sting 10.1.2. 5. Listing of rease<br>Patient ID | sons for tr | eatment d | iscontinua | ntion other the Reason | nan progres | | Specify | <u>.</u> |
| Tatient ID | | | | Reason | | | opeen, | |
| sting 10.1.2. 6. Listing of rea | sons for s | tudy diago | ntinuotion | other then | rogragiva | digagga | | |
| Patient ID | 50115 101 5 | iddy disco | Reas | | nogressive | Spec | eify | |
| | | | | | | - | | |
| | | | 1 | A.E.c | | | | |
| sting 10.1.2. 7. Listing of trea | atment dis | | on due to | AES. | | | | nificant |

## 10.1.3 Protocol deviations.

Listing 10.1.3. 1 Elegibility: Patients who entered the study even though they did not satisfy the entry criteria.

| Dose level | Patient id | I-E criteria no fulfilled | Deviation |
|---|---|---|---|
| sisting 10.1.3. 2 Protocol | l deviations: Patients de | eveloping withdrawal criteria but | were not |
| Daga lawal | Patient id | Deviatio | n |
| Dose level | 1 Wient iu | | |
| Listing 10.1.3. 3 Protocol | l deviations: Patients w | ho received incorrect dose or sch | |
| | | ho received incorrect dose or scho | |
| Listing 10.1.3. 3 Protocol Dose level | l deviations: Patients w Patient id | | n |

# 11 Appendix II. Efficacy evaluation.

## 11.1 Baseline characteristics.

# 11.1.1 Patients characteristics at baseline.

| | Total ( | N=XX) |
|------------------------------------|---------|-------|
| | N | % |
| Race: | | |
| Caucasian | | |
| Black | | |
| Other* | | |
| Age grouped: | | |
| 18 – XX years | | |
| XX – YY years | | |
| ≥ YY years | | |
| Patient id and race as a footnote. | | |

<sup>\*\*</sup> Stands for Not Applicable. Specify details in the footnote.

Table 11.1.1. 2. Summary statistics: baseline characteristics.

| | N | Missing | Median | Min | Max | Mean | SD |
|-------------|---|---------|--------|-----|-----|------|----|
| Age (years) | | | | | | | |
| Weight (Kg) | | | | | | | |

# 11.1.2 Histology and time from diagnosis.

Table 11.1.2. 1. Cancer diagnosis at baseline.

| Table 11.1.2. 1. Cancel diagnosis at basenile. | Tota | al (N=XX) |
|---|---|---|
| | N | % |
| Tumor type*: | | |
| Endometrial | | |
| Endometroid | | |
| Papillary Serous | | |
| Mixed | | |
| Clear cell | | |
| Other** | | |
| Cervix | | |
| Squamus cells carcinoma | | |
| Adenocarcinoma | | |
| Adenosquamus | | |
| Other** | | |
| Histology Grade: | | |
| Well differentiated | | |
| Moderately differentiated | | |
| Poorly differentiated | | |
| Undifferentiated | | |
| Unknown | | |
| Current Disease | | |
| Locally advanced | | |
| Metastatic | | |
| Number of Sites involved (target-non target): | | |
| 1 | | |
| 2 | | |
| 3 | | |
| > 3 | | |
| Summary Statistics of Number of Sites involved (target-non | | |
| target): | | |
| N | | |
| Median | | |
| Minimum | | |
| Maximum | | |

Programming Notes: Percentage is based on total patient included.

\* One table for each group. \*\* See listing 11.1.2.5

| | | | | <u>_</u> | N | % |
|---|---|---|---|---|---|---|
| IA | | | | | • | , , |
| IB | | | | | | |
| ••• | | | | | | |
| Table 11 1 2 3 | Sites for target and | l non-target legio | ne | | | |
| Sites | Sites for target and | i non-target resio | 115. | | | otal |
| Bone | | | | | N | % |
| Lung | | | | | | |
| Listing 11.1.2. 4 | 4. Listing of patien | t histology. | | | | |
| Patient ID | Tumor type<br>Stage | Histology Gr | ade . | ••••• | | Current s |
| | Stage | | | | | |
| Listing 11 1 2 5 | Ligting of all and | tum on tree | | | | |
| Patient ID | Listing of other : Histology | tumor types. | | | S | specify |
| I attent ID | ilistology | | ••••• | | ~ | peeny |
| | . Listing of target | | | • | | athod |
| Listing 11.1.2. 6 Patient ID | . Listing of target Target/non | | sions. Site/Subsit | e | M | ethod |
| Patient ID | Target/non | ı-target | Site/Subsit | e | М | ethod |
| Patient ID Listing 11.1.2. | Target/non 7. Listing of patien | a-target<br>ats with only one | Site/Subsit | | | |
| Patient ID | Target/non | ats with only one arget Site B | Site/Subsit | | | ethod<br>sly irradiate |
| Patient ID Listing 11.1.2. | Target/non 7. Listing of patien Target/non-ta | ats with only one arget Site B | Site/Subsit | | | |
| Patient ID Listing 11.1.2. Patient ID | Target/non 7. Listing of patien Target/non-ta | ats with only one arget Site B | Site/Subsit | N) | Previou | ısly irradiate |
| Patient ID Listing 11.1.2. 7 Patient ID Table 11.1.2. 8. | 7. Listing of patien Target/non-ta Histology/Cyt | ats with only one arget Site Brology | Site/Subsit | N) | Previou | ısly irradiate |
| Patient ID Listing 11.1.2. 7 Patient ID Table 11.1.2. 8. | 7. Listing of patien Target/non-ta Histology/Cyt Summary statistics | ats with only one arget Site Brology | single lesion. iopsy/FNA(Y/ | (N) | Previou<br>diagnosis and t | isly irradiate |
| Patient ID Listing 11.1.2. 7 Patient ID Table 11.1.2. 8. Time from f infusion (mo | 7. Listing of patien Target/non-ta Histology/Cyt Summary statistics irst diagnosis to onths) | ats with only one arget Site Brology s of cancer diagnomy first | single lesion. iopsy/FNA(Y/ | (N) | Previou<br>diagnosis and t | isly irradiate |
| Patient ID Listing 11.1.2. 7 Patient ID Table 11.1.2. 8. Time from f infusion (mo | 7. Listing of patien Target/non-ta Histology/Cyt Summary statistics irst diagnosis to onths) ast progression t | ats with only one arget Site Brology s of cancer diagnomy first | single lesion. iopsy/FNA(Y/ | (N) | Previou<br>diagnosis and t | isly irradiate |
| Patient ID Listing 11.1.2. 7 Patient ID Table 11.1.2. 8. Time from finfusion (more from 1 infusion (more f | 7. Listing of patien Target/non-ta Histology/Cyt Summary statistics irst diagnosis to onths) ast progression to onths) | ats with only one arget Site Brology s of cancer diagnomy first | single lesion. iopsy/FNA(Y/ | (N) | Previou<br>diagnosis and t | isly irradiat |
| Patient ID Listing 11.1.2. 7 Patient ID Table 11.1.2. 8. Time from finfusion (more from 1 infusion (more f | 7. Listing of patien Target/non-ta Histology/Cyt Summary statistics irst diagnosis to onths) ast progression t | ats with only one arget Site Brology s of cancer diagnomy first | single lesion. iopsy/FNA(Y/ | (N) | Previou<br>diagnosis and t | isly irradiate |
| Patient ID Listing 11.1.2. 7 Patient ID Table 11.1.2. 8. Time from f infusion (more from l infusion (more) (*) SD stands | 7. Listing of patien Target/non-ta Histology/Cyt Summary statistics irst diagnosis to onths) ast progression to onths) | ats with only one arget Site Brology s of cancer diagnor N first to fir | single lesion. iopsy/FNA(Y/ | (N) | Previou<br>diagnosis and t | isly irradiate |
| Patient ID Listing 11.1.2. 7 Patient ID Table 11.1.2. 8. Time from f infusion (more from l infusion (more) (*) SD stands | Target/non 7. Listing of patien Target/non-ta Histology/Cyt Summary statistics irst diagnosis to onths) ast progression to onths) for standard dev anticancer thera | ats with only one arget Site Brology s of cancer diagnor N first to fir | single lesion. iopsy/FNA(Y/ | Time from Min | Previou<br>diagnosis and t | isly irradiate |

Table 11.1.3. 2 Radiotherapy type. Total (N=XX) **%** External Brachytherapy **IORT** Table 11.1.3. 3 Radiotherapy setting Total (N=XX) **%** N Radiotherapy Chemoradiotherapy Listing 11.1.3. 4 Patients with prior radiotherapy Site **Type** Setting **First Patient ID** Last date date Listing 11.1.3. 5 Patients with prior surgery. **Patient ID** Intention **Site and Procedures** Residual diseas **Date** Table 11.1.3. 6 Summary statistics of prior systemic anticancer therapy. Median Min Max Mean SD No of lines No of agents Table 11.1.3. 7 Number of lines and agents of systemic anticancer therapy. Total (N=XX) **%** Number of lines 2 3 > 3 Number agents 1 2 3 > 3 Table 11.1.3. 8 Prior anticancer agents. Antineoplastic and Immunomodulating agents N **%** (ATC-clas. Levels 1-4) Antineoplastic Agents (L01) Endocrine therapy (L02)

# 11.1.4 Prior history.

| Listing 11.1.4. 1. Prior history | Listing | 11. | 1.4. | 1. I | Prior | history |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

| Listing 11.1.4. 1. Pr | | D | 0 | Danaharah da 4 |
|---|---|---|---|---|
| Patient ID. | | Description | Onset dat | Resolved date |
| 11.1.5 Physical | l examination, vital | signs, electroca | rdiogram and other tests. | |
| Table 11.1.5. 1 Phy | ysical examination at b | aseline. | | |
| | | | Total (N= | XX) |
| | | | N | % |
| Physical Exan | nination: | | | |
| Normal | | | | |
| Abnormal | | | | |
| <b>ECOG-PS:</b> | | | | |
| 0 | | | | |
| 1 | | | | |
| ECG: | | | | |
| Normal | | | | |
| Abnormal | | | | |
| LVEF | | | | |
| Normal | | | | |
| Abnormal | 1 4 1 | | | |
| Adequate birt<br>Yes | in control: | | | |
| No | | | | |
| NA* | | | | |
| Pregnancy tes | · <b>+</b> | | | |
| Positive | ot . | | | |
| Negative | | | | |
| | "Not applicable" | | | |
| 1 VI Stands 101 | 110t applicable | | | |
| Listing 11.1.5. 2 L | isting of abnormal ECO | J. | | |
| Patient ID | <u> </u> | ECG result | | Specify |
| - ************************************* | | | | эрссау |
| Listing 11.1.5. 3 L | isting of LVEF. | | | |
| Patient ID | LVEF(%) | Method | Institutional normal rai | nge Resu |

| | N | Missing | Median | Min | Max | Mean | SD |
|------------------------|---|---------|--------|-----|-----|------|----|
| Heart Rate (beats/min) | | | | | | | |
| BPS (mmHg) | | | | | | | |
| BPD (mmHg) | | | | | | | |
| Temperature (°C) | | | | | | | |

# 11.1.6 Hematological values at baseline.

Table 11.1.6. 1. Hematological abnormalities at baseline.

| | Gr | ade 1 | Gra | ide 2 | Gra | de 3 | Gra | Grade 4 | | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| _ | N | % | N | % | N | % | N | % | N | % |
| Leukopenia | | | | | | | | | | |
| Neutropenia | | | | | | | | | | |
| Anemia | | | | | | | | | | |
| Thrombocytopenia | | | | | | | | | | |
| Lymphopenia | | | | | | | | | | |

Table 11.1.6. 2. Hematology at baseline. Last value before treatment.

| | N | Missing | Median | Min | Max | Mean | SD |
|-------------|---|---------|--------|-----|-----|------|----|
| Leukocytes | | | | | | | |
| Neutrophils | | | | | | | |
| Hemoglobin | | | | | | | |
| Platelets | | | | | | | |
| Lymphocytes | | | | | | | |

Listing 11.1.6. 3. Hematology at baseline. Patients with hematological parameters missing.

| Patient ID. | Exam |
|-------------|------|

Listing 11.1.6. 4. Hematology at baseline. Abnormalities grade >=2.

| Patient ID. | Parameter | Value | Grade |
|-------------|-----------|-------|-------|

# 11.1.7 Biochemical values at baseline

Table 11.1.7. 1. Biochemical abnormalities at baseline.

| | Gi | Grade I | | iae 2 | Gra | iae 3 | Gra | iae 4 | 10 | 1 otai |
|-----|----|---------|---|-------|-----|-------|-----|-------|----|--------|
| | N | % | N | % | N | % | N | % | N | % |
| AST | | | | | | | | | | |
| ALT | | | | | | | | | | |

Direct Bilirubin

Total Bilirubin

Table 11.1.7. 2. Biochemistry at baseline. Last value before treatment.

| | N | Missing | Median | Min | Max | Mean | Max |
|------------------|---|---------|--------|-----|-----|------|-----|
| AST | | | | | | | |
| ALT | | | | | | | |
| Total Bilirubin | | | | | | | |
| Direct Bilirubin | | | | | | | |

| Patient ID | <u>, </u> | | | | Exam | | | | - | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Listino 11 1 7 | 4. Biochemistr | v at hase | line Ahn | ormaliti | es orade >= | 2 | | | • | | |
| Patient ID | | | Parame | | es grade - | Value | | | Grade | | |
| | er metabolic | | | | | | | | | | |
| Table 11.1.8. | 1. Other metabo | olic abno<br><b>Grade</b> | | at baseli<br>Grad | | Grad | de 3 | Gra | ade 4 | To | otal |
| | | | % | N | % | N | % | N | % | N | ( |
| Hyperglyc | emia | | | | | | | | | | |
| * All metab<br>Table 11.1.8. | olic paramete 2. Other metabo | ers susc | eptible t | to be grat baseli | raded as p | oer NCI<br>Hypo). La | -CTCAE ast value be | v3.0<br>fore treat | tment. | | |
| | | N | Miss | ing | Median | M | in I | Max | Mean | | SD |
| Glucose * | | | | | | | | | | | |
| Patient ID | . 3. Patients with | h metabo | lic param | eters mis | | | | | | | |
| Patient ID | . 4. Other metal | | oaseline. A | Exa | m<br>alities grade | >=2. | | Value | | Gra | ade |
| Patient ID Listing 11.1.8 Patient ID 11.1.9 Sign Table 11.1.9.1 | . 4. Other metal | bolic at b | paseline. A | Exa Abnorma Param | ulities grade neter | | nde 3 | | ade 4<br>% | | ade<br>otal |
| Patient ID Listing 11.1.8 Patient ID 11.1.9 Sign Table 11.1.9.1 SOC/Medlterm General | . 4. Other metal . and sympto . Summary stati DRA Preferr Abdominal Distension | bolic at b<br>oms at b<br>istics: Sig<br>Gr | paseline. A paseline. gns and syrade 1 | Exa Abnorma Param /mptoms Gr | and alities grade neter | Gra | | Gr | | To | otal |
| Listing 11.1.8 Patient ID 11.1.9 Sign Table 11.1.9.1 SOC/Mediterm General Disorders Pain | . 4. Other metal . and sympto . Summary stati DRA Preferr Abdominal Distension | oms at b | paseline. A paseline. gns and syrade 1 % | Exa Abnorma Param /mptoms Gr N | and additional state of the sta | Gra | | Gr | | To | otal |
| Listing 11.1.8 Patient ID 11.1.9 Sign Table 11.1.9.1 SOC/Mediterm General Disorders Pain | . 4. Other metalo. as and sympto Summary stati DRA Preferro Abdominal Distension | oms at b | paseline. A paseline. gns and sy pade 1 % | Exa Abnorma Param /mptoms Gr N | alities grade neter s. rade 2 % | Gra | | Gr.<br>N | | To<br>N | otal |
| Listing 11.1.8 Patient ID 11.1.9 Sign Table 11.1.9.1 SOC/Medl term General Disorders Pain Table 11.1.9.2 (*) SD stand | . 4. Other metalo. as and sympto Summary stati DRA Preferro Abdominal Distension | oms at be istics: Signature of the istics: Sig | paseline. A paseli | Abnorma Param /mptoms Gr N | alities grade neter s. cade 2 % | Gra<br>N | 9/0 | Gr.<br>N | 9/0 | To<br>N | otal |

# 11.1.10 Concomitant therapy.

| | nedication (AT | nt therapy started at b | baseline. | | | |
|---|---|---|---|---|---|---|
| (ATC level 1) | (ATC lev | · | | N | | % |
| | ( | / | | | | |
| Гable 11.1.10.2. С | oncomitant medicat | ion characteristics at | haseline. | | | |
| | | | | Total ( | N=XX) | |
| | | | N | • | % | |
| Number of Syst | tems (ATC1) | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| 3<br>> 3 | | | | | | |
| Number of ager | nts (ATC4) | | | | | |
| 1 | 115 (11101) | | | | | |
| 2<br>3 | | | | | | |
| > 3 | | | | | | |
| T.1.1. 11 1 10 2 C | | -44-1-4-1 | | C | | |
| 1able 11.1.10.3. C | oncomitant therapy N | started at baseline. Su <b>Median</b> | Min | Max | Mean | SD; |
| | 11 | Median | IVIIII | Max | Mean | SD |
| Table 11.1.10. 4. С | oncomitant therapy N | started at baseline. Su Median | ummary of number | er of agents inv Max | wolved (ATC4). Mean | SD* |
| Listing 11.1.10. 5. 1 | Listing of Baseline of | characteristics: Conco | omitant therapy. | | | |
| Patient ID | Start date | ATC code | Route | I | Reason for use | _<br>_ |
| | | | | | | _<br>_ |
| 11.2 Eec. | | | | | | |
| 11.2 Efficacy. | | | | | | |
| 11.2.1 Response | 2. | | | | | |
| Listing 11.2.1. 1. Lis | sting of patients excl | luded from the efficac | cy analysis. | | | |
| Patient ID | • | | Reason | | | |
| Table 11.2.1. 2. Pati | ients evaluable for e | fficacy. | | | | |
| Evaluable | | | | Total (N: | =XX) | |
| | | | N | | % | |
| Yes | | | | | | _ |
| No<br>Total | | | | | | |

Table 11.2.1. 3. Best response in all evaluable patients.

| Response | N | % | CI (95%) |
|----------------------------|---|---|----------|
| Complete Response (CR) | | | |
| Partial Response (PR) | | | |
| Stable Disease ≥ 4 months* | | | |
| Stable Disease (SD) | | | |
| Progression Disease (PD)** | | | |

Programming Notes: Percentage is based on the total of patient evaluable for efficacy

- (\*) Patients who are free from progression in the tumor evaluation at 4 months
- (\*\*) Patients with Early PD will also be included in this category (provided that they receive at least two infusions of PM00104)

NOTE: An analysis of best response in the 10 and 18 first evaluable patients in the group 1 and group 2 respectively will also be performed. Table 11.2.1.3 will be repeated at this interim analysis and at the end of the study.

Table 11.2.1. 4. Best response in all treated patients.

| Response | N | % | CI (95%) |
|----------------------------|---|---|----------|
| Complete Response (CR) | | | |
| Partial Response (PR) | | | |
| Stable Disease ≥ 4 months* | | | |
| Stable Disease (SD) | | | |
| Progression Disease (PD)** | | | |
| Not evaluable | | | |

Programming Notes: Percentage is based on total patient of patients treated (\*)Patients who are free from progression in the tumor evaluation at 4 months

(\*\*) Patients with Early PD will also be included in this category (provided that they receive at least two infusions of PM00104)

Table 11.2.1. 5. Progression Free Survival status at 4 months (PFS4) in all evaluable patients.

| PFS4 | Total | (N=XX) |
|-------------|-------|------------|
| FF 54 | N | % (95% CI) |
| Yes | | |
| No | | |
| No<br>Total | | |

Table 11.2.1. 6. Progression Free Survival status at 4 months (PFS4) in all treated patients.

| PFS4 | Total | (N=XX) |
|-------|-------------------------|------------|
| FF 54 | $\overline{\mathbf{N}}$ | % (95% CI) |
| Yes | | |
| No | | |
| Total | | |

Table 11.2.1. 7. Progression Free Survival status at 6 months (PFS6) in all evaluable patients.

| PFS6 | Total | l (N=XX) |
|-------|-------------------------|------------|
| FF30 | $\overline{\mathbf{N}}$ | % (95% CI) |
| Yes | | |
| No | | |
| Total | | |

| Table 11.2.1. 8. | Progression Free | Survival status at 6 mo | nths (PFS6) in al | I treated patients. |
|---|---|---|---|---|

| PFS6 | Total | l (N=XX) |
|-------|-------|------------|
| rrso | N | % (95% CI) |
| Yes | | |
| No | | |
| Total | | |

#### 11.2.2 Time-to-event variables.

#### Table 11.2.2. 1. Duration of response.

**Summary** 

N=XX

Events X (XX.X%)

Censored X (XX.X%)

Median X.X 95% CI (X.X-X.X)

DR > 3 months XX.X% 95% CI XX.XX%-XX.X%)

DR > 6 months XX.X% 95% CI XX.XX%-XX.X%)

# Table 11.2.2. 2. Progression Free Survival (Kaplan-Meier estimates in all evaluable patients).

**Summary** 

N=XX

Events X (XX.X%)

Censored X (XX.X%)

Median X.X 95% CI (X.X-X.X)

PFS rate at 4 months XX.X% 95% CI XX.XX%-XX.X%)

PFS rate at 6 months XX.X% 95% CI XX.XX%-XX.X%)

#### Table 11.2.2. 3. Progression Free Survival (Kaplan-Meier estimates in all treated patients).

Summary

N=XX

Events X (XX.X%)

Censored X (XX.X%)

Median X.X 95% CI (X.X-X.X)

PFS rate at 4 months XX.X% 95% CI XX.XX%-XX.X%)

PFS rate at 6 months XX.X% 95% CI XX.XX%-XX.X%)

# Table 11.2.2. 4. Overall Survival. Evaluable population.

**Summary** 

N=XX

Events X (XX.X%)

Censored X (XX.X%)

Median X.X 95% CI (X.X-X.X)

OS rate at 6 months XX.X% 95% CI XX.XX%-XX.X%)

OS rate at 12 months XX.X% 95% CI XX.XX%-XX.X%)

| Summary<br>N=XX | | | | | | |
|---|---|---|---|---|---|---|
| Events X (XX | .X%) | | | | | |
| Censored X (2 | , | | | | | |
| Median X.X 9 | | | <b>3/ 3/3/0/ 3/3/ 3/0/</b> ) | | | |
| | | | X.XX%-XX.X%)<br>XX.XX%-XX.X% | ` | | |
| OS Tate at 12 | months AA.A | 70 73 70 C1 2 | AA,AA /0-AA,A /0 | <i>)</i> | | |
| Table 11.2.2. 6. Fo | ollow-up period. | | | | | |
| Parameter | Medi | an 95 | % CI Lower boun | d 95° | % CI Upj | per bou |
| PFS | | | | | | |
| OS | | | | | | |
| 11.2.3 Patients | s with clinical b | enefit. | | | | |
| Listing 11.2.3. 1. C | Characteristics of p | atients with cli | nical benefit*. | | | |
| | naracteristics | | Outcome prior trea | ntment | | PM00104 |
| treatment | (DC 171 ) I | 710 T | | | | C DE |
| Patient Sex/Ag | ge/PS Histolo | gy N° Prio | r Last prior Cyc | les B | est TTP | Cyc PFS |
| 08 | | CT Line | s Treatment recei | ived Res | nonse | |
| | | CT Eme | 3 Treatment rece | ived ites | ponse | |
| (*) Clinical ben | efit defined as | patients who | experience any of | the follo | wing CR | or PR or PFS |
| | | • | | the follo | wing CR ( | or PR or PFS |
| | efit defined as | • | | the follo | wing CR o | or PR or PFS |
| | marker evolutio | on/response ( | | the follo | wing CR ( | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4. 1 C. | marker evolutio | on/response (<br>ummary. | group 1). | the follo | wing CR ( | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4. 1 C. | marker evolution so | on/response (<br>ummary. | group 1). | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4.1 C. N Median | marker evolution so | on/response (<br>ummary. | group 1). | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4.1 C. N Median Max | marker evolution so | on/response (<br>ummary. | group 1). | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4.1 C. N Median | marker evolution so | on/response (<br>ummary. | group 1). | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4. 1 C. N Median Max Min | marker evolution so Baselin | on/response ( ummary. e Cyc 1 | Cyc 2 | | | or PR or PFS |
| Table 11.2.4. 1 C. N Median Max Min Table 11.2.4. 2 C. | marker evolution so Baselin A-125 evolution d | on/response ( ummary. ne Cyc 1 uring treatment | Cyc 2 C | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4. 1 C. N Median Max Min | marker evolution so Baselin | on/response ( ummary. e Cyc 1 | Cyc 2 | | | or PR or PFS |
| Table 11.2.4. 1 C. N Median Max Min Table 11.2.4. 2 C. | marker evolution so Baselin A-125 evolution d | on/response ( ummary. ne Cyc 1 uring treatment | Cyc 2 C | | | or PR or PFS |
| Table 11.2.4. 1 C. N Median Max Min Table 11.2.4. 2 C. Patient ID | marker evolution so Baselin A-125 evolution d | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 | Cyc 2 C | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4.1 C. N Median Max Min Table 11.2.4.2 C. Patient ID | Marker evolution so Baselin A-125 evolution d Baseline III. Safety eva | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 | Cyc 2 C | | | or PR or PFS |
| Table 11.2.4. 1 C. N Median Max Min Table 11.2.4. 2 C. Patient ID | Marker evolution so Baselin A-125 evolution d Baseline III. Safety eva | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 | Cyc 2 C | | | or PR or PF |
| 11.2.4 Tumor Table 11.2.4.1 C. N Median Max Min Table 11.2.4.2 C. Patient ID 12 Appendix 12.1 Extent o | Marker evolution so A-125 evolution so Baselin A-125 evolution d Baseline III. Safety evaluation description | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 aluation. | Cyc 2 C | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4.1 C. N Median Max Min Table 11.2.4.2 C. Patient ID 12 Appendix 12.1 Extent o | Marker evolution so Baselin A-125 evolution d Baseline III. Safety eva | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 aluation. | Cyc 2 C | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4.1 C. N Median Max Min Table 11.2.4.2 C. Patient ID 12 Appendix 12.1 Extent o 12.1.1 Treatm | Marker evolution so A-125 evolution so Baseline A-125 evolution d Baseline III. Safety eva f exposure. ent administrat | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 aluation. | Cyc 2 C | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4. 1 C. N Median Max Min Table 11.2.4. 2 C. Patient ID 12 Appendix 12.1 Extent o 12.1.1 Treatm Table 12.1.1. 1. Cy | Marker evolution state A-125 evolution state Baselin A-125 evolution d Baseline III. Safety evaluation d f exposure. ent administrate celes administered. | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 aluation. | Cyc 2 C | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4.1 C. N Median Max Min Table 11.2.4.2 C. Patient ID 12 Appendix 12.1 Extent o 12.1.1 Treatm | Marker evolution state A-125 evolution state Baselin A-125 evolution d Baseline III. Safety evaluation d f exposure. ent administrate celes administered. | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 aluation. | Cyc 2 C | | | or PR or PFS |
| 11.2.4 Tumor Table 11.2.4. 1 C. N Median Max Min Table 11.2.4. 2 C. Patient ID 12 Appendix 12.1 Extent o 12.1.1 Treatm Table 12.1.1. 1. Cy | Marker evolution state A-125 evolution state Baselin A-125 evolution d Baseline III. Safety evaluation d f exposure. ent administrate celes administered. | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 aluation. | Cyc 2 Company of the per patient. Cycle 2 | | | |
| 11.2.4 Tumor Table 11.2.4.1 C. N Median Max Min Table 11.2.4.2 C. Patient ID 12 Appendix 12.1 Extent o 12.1.1 Treatm Table 12.1.1.1. Cy Cycles per pa | Marker evolution state A-125 evolution state Baselin A-125 evolution d Baseline III. Safety evaluation d f exposure. ent administrate celes administered. | on/response ( ummary. ne Cyc 1 uring treatment Cycle 1 aluation. | Cyc 2 Company of the per patient. Cycle 2 | | | |

Table 12.1.1. 2. Summary of cycles administered.

| Table 12.1.1. 2. Summary of cycles admin | istered. | | | | |
|---|---|---|---|---|---|
| N | Median | Min | Max | Mean | SD* |
| (*) SD stands for standard deviatio | n | | | | |
| Table 12.1.1. 3. Dose intensity. | | | | | |
| | N | Median | Min Min | | Max |
| Cumulative dose (mg/ m²) | | | | | |
| Treatment duration (wk) | | | | | |
| Dose intensity (mg/m² wk) | | | | | |
| Relative dose intensity (%) | | | | | |
| 12.1.2 Dose delays. Table 12.1.2. 1. Dose delay. | | | | | |
| | | N | | | % |
| Number of patients treated | | | | | |
| Number of patients with any dose | delay | | | | |
| Number of cycles administered | | | | | |
| Number of cycles susceptible to b | e delayed | | | | |
| Patients with | | | | | |
| No delays | | | | | |
| 1 cycle delayed | | | | | |
| 2 cycles delayed | | | | | |
| ≥ 3 cycles delayed | 1 1 | | | | |
| Number of cycles with dose de | lay* | | | | |

Programming Notes: Percentage is based on number of cycle susceptible to be delayed.

Table 12.1.2. 2. Dose delay according to their relationship to study drug.

| , , , | Treatment related** | | Non – Treat | ment related |
|---|---|---|---|---|
| | N | % | N | % |
| Patients with | | | | |
| No delays | | | | |
| 1 cycle delayed | | | | |
| 2 cycles delayed | | | | |
| ≥ 3 cycles delayed | | | | |
| Number of cycles with dosing delay | | | | |

# Programming Notes:

- \* Denominator = Number of cycles susceptible to be delayed. \*\* Hematological reason / Non hematological reason.

<sup>\*</sup> Denominator = Number of cycles susceptible to be delayed.

Table 12.1.2. 3. Length of dose delay.

| | Treatmen | Treatment related* Non – Treatment relate | | | | Total |
|---|---|---|---|---|---|---|
| | N | % | N | % | N | % |
| Lenght of delay | | | | | | |
| 1-7 days | | | | | | |
| 7 – 14 days | | | | | | |
| > 14 days | | | | | | |

## Programming Notes:

- \* Denominator = Number of cycles susceptible to be delayed.
- \*\* Hematological reason / Non hematological reason.

Table 12.1.2. 4 . Dose delay and reason by cycle.

| Cyc | ele 2 | Cy | cle 3 | • • | | To | tal |
|-----|-------|----|-------|-----|---|----|-----|
| N | % | N | % | N | % | N | % |

Number of delays

Treatment related\*

Hematological reason

Non hematological reason

Non Treatment related\*

Programming Notes: \* Denominator = Number of cycles susceptible to be delayed.

Listing 12.1.2. 5. Listing of patient with dose delay.

| Patient II | Cycle | Reason of delay | Comments | Delay (days) |
|------------|-------|-----------------|----------|--------------|

#### 12.1.3 Dose reduction.

Note: All dose reductions will be considered and described, specifying the reason for reduction (hematological toxicity, non hematological toxicity or other causes not due to study drug).

Table 12.1.3. 1 Dose reduction.

| | N | % |
|--------------------------------------|---|---|
| Number of patients treated | | |
| Number of patients with dose reduced | | |
| Number of cycles administered | | |
| Patients with | | |
| Nº reductions | | |
| 1 cycle reduction | | |
| 2 cycle reductions | | |
| ≥ 3 cycle reductions | | |
| Number of cycles with dose reduction | | |

Programming Notes: Percentage is based on number of cycle susceptible to be reduced.

Table 12.1.3. 2 Dose reduction according to their relationship to study drug.

| | Treatmen | t related** | Non – Treat | ment related |
|----------------|----------|-------------|-------------|--------------|
| | N | % | N | % |
| Patients with | | | | |
| N° reductions | | | | |
| 1 reduction | | | | |
| 2 reductions | | | | |
| ≥ 3 reductions | | | | |

Number of cycles with dose reduction\*

Programming Notes:\* Denominator = Number of cycles susceptible to be reduced.

\*\* Hematological reason / Non-hematological reason.

Table 12.1.3. 3 Dose reduction and reason by cycle.

| | Cycle 2 | | Cycle 3 | | ••• | | Total | |
|--------------------------|---------|---|---------|---|-----|---|-------|---|
| _ | N | % | N | % | N | % | N | % |
| Number of patients | | | | | | | | |
| Number of delays | | | | | | | | |
| Treatment related* | | | | | | | | |
| Hematological reason | | | | | | | | |
| Non hematological reason | | | | | | | | |
| Non Treatment related* | | | | | | | | |

Programming Notes:\* Denominator = Number of cycles susceptible to be reduced.

Listing 12.1.3.4 Patient with dose reduction.

| Patient ID | Cycle Reason of reduction | Comments | Reduction (%) |
|-------------------|-------------------------------|----------|---------------|
| 12.1.4 Skippe | ed doses. | | |
| Table 12.1.4. 1 S | kipped doses. | | |
| | | N | % |
| Number of pat | ients treated with at least 2 | | |
| infusions | | | |
| Number of pat | ients with any skipped dos | | |
| Number of pat | ients with any skipped dos | | |
| (drug related) | | | |
| Number of cyc | cles administered | | |
| Number of cyc | cles susceptible to have any | | |
| omission | 1 | | |
| Number of cyc | eles with at least one skipp | | |
| dose (drug rela | | | |
| Day 8 | , | | |
| Day 15 | | | |
| Day 8+15 | | | |

| | Tre | eatment related** | Non – Treatment related | |
|---|---|---|---|---|
| | N | %(of all cycles) | N | %(of all cycles) |
| Day 8 | | | | |
| Day 15 | | | | |
| Day 8+15 | | | | |

Listing 12.1.4.3. Listing of patients with skipped doses.

| Patient ID | Cycle/infusion (skipped dose) | Reason (drug related/other) | Comments |
|---|---|---|---|

## 12.2 Toxicity.

# 12.2.1 Adverse events.

- Table 12.2. 1 Drug related adverse events. Worst case per patient.
- Table 12.2. 2 Drug related adverse events occurring in > 10% of all patients. Worst case per patient.
- Table 12.2. 3 All adverse events regardless relationship. Worst case per patient.
- Table 12.2.4 All adverse events regardless relationship occurring in > 10% of all patients. Worst case per patient.
- Table 12.2. 5 Drug related adverse events. Worst case per cycle.
- Table 12.2. 6 Drug related adverse events occurring in > 10% of all cycles. Worst case per cycle.
- Table 12.2. 7 All adverse events regardless relationship. Worst case per cycle.
- Table 12.2. 8 All adverse events regardless relationship occurring in > 10% of all cycles. Worst case per cycle.

| System Organ Class/<br>Preferred Term | Gr | ade 1 | Gra | ade 2 | Gra | ade 3 | Gra | de 4 | Т | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | % | N | % | N | % | N | % | N | % |
| System Organ Class 1 Preferred Term | | | | | | | | | | |
| System Organ Class 2 Preferred Term | | | | | | | | | | |

<sup>\*</sup> Percentages are based on the safety population. Table shows number of distinct patients with events.

#### 12.2.2 Serious toxicity rate.

Table 12.2.2. 1 Serious toxicity rate by group

| | Gro | up XX |
|-----|-----|-------|
| | N | % (*) |
| Yes | | |
| No | | |

<sup>(\*)</sup> Based on the first 10 consecutive patients by group.

Listing 12.2.2. 1 Listing of patients with any serious toxicity rate (grades 3-4) by group.

| <b>Patient ID</b> | MedDRA | Crada | Relation with | | Ongot data | End Data |
|---|---|---|---|---|---|---|
| Patient ID | preferred term | Grade | the study drug | ••••• | Onset date | End Date |

#### 12.2.3 Serious adverse events.

All serious adverse events will be listed only for the purpose of reconciliation with the database of pharmacovigilance. The listings provided by the Product Safety department will be used for the clinical study report.

Listing 12.2.3. 1. Listing of SAEs

| Patient ID | MedDRA<br>preferred term | Grade | Relation with the study drug | •••• | Start date | End Date |
|---|---|---|---|---|---|---|
| Listing 12.2.3 | 2. Listing of deaths r | elated to study d | lnıg | | | |
| Patient ID | Cause of Des | | om last infusion | Auto<br>(Y/N | | psy report<br>able (Y/N) |

# 12.3 Laboratory evaluation.

## 12.3.1 Hematological abnormalities.

Table 12.3.1. 1 Hematology worst grade per patient.

| | Gra | Grade 1 | | Grade 2 | | Grade 3 | | Grade 4 | | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | % | N | % | N | % | N | % | N | % |
| Leukopenia<br>Neutropenia | | | | | | | | | | |

Anemia

Thrombocytopenia Lymphopenia

Programming Notes: Percentages are based on the safety population.

Table 12.3.1. 2 Hematology worst grade per cycle.

| Grade 1 | | Gra | Grade 2 | | Grade 3 | | Grade 4 | | Total |
|---|---|---|---|---|---|---|---|---|---|
| <br>N | <b>%</b> | N | <b>%</b> | N | % | N | % | N | % |

Leukopenia

Neutropenia

Anemia

Thrombocytopenia

Lymphopenia

Programming Notes: Percentages are based on the safety population.

Supportive listing: Patients with any hematological abnormalities grade 3-4.

| CICIE VS.0 | Patient | Lab. test | Cycle | Examination dat | N | Std. value | xLLN | Grade NCI<br>CTCAE v3.0 |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

| Listing 12.3.1. 4 | Listing of patients | with haematology evaluations missing. |
|---|---|---|
| Patient | Cycle | Lab. test |

Table 12.3.1. 5 Time course and recovery from hematological toxicities.

| | N | All c | ycles |
|----------------------------------------|---|--------|-------|
| | N | Median | Range |
| Neutrophils | | | |
| Day of nadir neutrophils count | | | |
| Nadir of neutrophils count (/mm3) | | | |
| Day of neutropenia G3-4 onset | | | |
| Day of recovery to grade ≤2 | | | |
| N° of days with grade 3-4 neutropenia | | | |
| Day of recovery to grade $\leq 1$ | | | |
| Platelets | | | |
| Day of nadir platelets count | | | |
| Nadir of platelets count (/mm3) | | | |
| Day of thrombopenia G3-4 onset | | | |
| Day of recovery to grade ≤2 | | | |
| N° of days with grade 3-4 thrombopenia | | | |
| Day of recovery to grade $\leq 1$ | | | |

Programming notes: (\*)Denominator = N of patients with Grade 3-4

Table 12.3.1. 6 Baseline grade and evolution of hematological toxicities.

| | Worst grade per patient | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Gra | de 0- | Gra | ide 2 | Grade 3 | | Gr | ade 4 |
| | N | <b>%</b> | N | <b>%</b> | N | <b>%</b> | N | <b>%</b> |
| Anemia (Baseline) | | | | | | | | |
| Grade 0-1 | | | | | | | | |
| Grade 2 | | | | | | | | |
| Grade 3 | | | | | | | | |
| Grade 4 | | | | | | | | |
| Neutropenia (Baseline) | | | | | | | | |
| Grade 0-1 | | | | | | | | |
| Grade 2 | | | | | | | | |
| Grade 3 | | | | | | | | |
| Grade 4 | | | | | | | | |
| Grade 0-1 | | | | | | | | |
| Grade 2 | | | | | | | | |
| Grade 3 | | | | | | | | |
| Grade 4 | | | | | | | | |

# 12.3.2 Biochemistry abnormalities.

Table 12.3.2. 1 Biochemistry worst grade per patient.

| Table 12.3.2. 1 Blochen | nsuy woi | st grade p | er patient. | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Grade 1 | | Gra | Grade 2 | | Grade 3 | | Grade 4 | | Total |
| | N | % | N | % | N | % | N | % | N | % |
| AST | | | | | | | | | | |
| ALT | | | | | | | | | | |
| Total Bilirubin | | | | | | | | | | |
| Direct Bilirubin | | | | | | | | | | |

Programming Notes: Percentages are based on the safety population.

Table 12.3.2. 2 Biochemistry worst grade per cycle.

| | Gr | Grade 1 | | Grade 2 | | Grade 3 | | Grade 4 | | Total |
|-----|----|---------|---|---------|---|---------|---|---------|---|-------|
| | N | % | N | % | N | % | N | % | N | % |
| AST | | | | | | | | | | |
| ALT | | | | | | | | | | |

Total Bilirubin

Direct Bilirubin

....

Programming Notes: Percentages are based on the safety population.

Table 12.3.2. 3 Supportive listing: Patients with any Biochemistry abnormalities grades 3-4.

| Patient ID | Lab. test | Cycle | Examination<br>date | N | Std. valı | xLLN | Grade |
|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|

Table 12.3.2. 5 Time course and recovery from biochemistry toxicities.

| N | All cycles | |
|---|------------|-------|
| N | Median | Range |

ALT

Day of peak ALT count

Nadir of ALT count (/mm3)

Day of ALT G3-4 onset

Day of recovery to grade ≤2

N° of days with grade 3-4 ALT increase

Day of recovery to grade  $\leq 1$ 

AST

Day of peak AST count

Nadir of AST count (/mm3)

Day of AST G3-4 onset

Day of recovery to grade ≤2

N° of days with grade 3-4 AST increase

Day of recovery to grade  $\leq 1$ 

Programming notes: (\*) Denominator= N of patients with Grade 3-4.

| Table 12.3.2. 6 | Baseline 9 | $\mathbf{g}$ rade and $\epsilon$ | evolution ( | of Biochemi | cal toxicities. |
|---|---|---|---|---|---|

| | | Worst grade per patient | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Grad | e 0-1 | Grade 2 | | Grade 3 | | Grade 4 | |
| | N | <b>%</b> | N | <b>%</b> | N | <b>%</b> | N | % |
| ALT (Baseline) | | | | | | | | |
| Grade 0-1 | | | | | | | | |
| Grade 2 | | | | | | | | |
| Grade 3 | | | | | | | | |
| Grade 4 | | | | | | | | |
| AST (Baseline) | | | | | | | | |
| Grade 0-1 | | | | | | | | |
| Grade 2 | | | | | | | | |
| Grade 3 | | | | | | | | |
| Grade 4 | | | | | | | | |
| Grade 0-1 | | | | | | | | |
| Grade 2 | | | | | | | | |
| Grade 3 | | | | | | | | |
| Grade 4 | | | | | | | | |

#### 12.3.3 Other metabolic abnormalities.

Table 12.3.3. 7 Metabolic abnormalities worst grade per patient.

| | | | Gra | Grade 1 | | Grade 2 | | Grade 3 | | Grade 4 | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | N | % | N | % | N | % | N | % | N | % |
| TT | 1 | • | | | | | | | | | | |

Hyperglycemia

• • • •

Table 12.3.3. 8 Metabolic abnormalities grade per cycle.

| _ | Gr | ade 1 | Grade 2 | | Grade 3 | | Grade 4 | | Total | |
|---|----|-------|---------|---|---------|---|---------|---|-------|---|
| | N | % | N | % | N | % | N | % | N | % |

Hyperglycemia

. . . .

Table 12.3.3. 9 Supportive listing: Patients with any metabolic abnormalities grades 3-4.

| Patient ID | Lab. test | Cycle | Examination date | N | Std. value | xLLN | Grade |
|---|---|---|---|---|---|---|---|

| T : .: 10 0 0 10 | T | 1 11 1 1 1 |
|---|---|---|
| $1 \cdot 1 \cdot$ | Listing of patients with met | abolic evaluations missing |
| Listing 12.3.3. 10 | Listing of patients with filet | abone evaluations imponing. |

| Patient | Cycle | Lab. test |
|---------|-------|-----------|

<sup>\*</sup> All metabolic parameters susceptible to be graded as per NCI-CTCAE v3.0

<sup>\*</sup> All metabolic parameters susceptible to be graded as per NCI-CTCAE v3.0

# 12.4 Vital Signs.

| signs. |
|--------|

| Vital Signs | Baseline | Cycle 1 | Cycle 2 | ••• | Cycle (X) |
|---|---|---|---|---|---|
| PS | | | | | |
| Weigth (Kg) | | | | | |
| LVEF (%) | | | | | |
| Table 12.4. 2 Listin | ng of abnormal ECC | <u>.</u> | | | |
| Patient id | Result | | S | Specify | |

# 12.5 Concomitant medication during treatment.

Table 12.5.1. 1. Agents of Concomitant therapy started during treatment.

| Concomitant medication (ATC1/ATC4) | | | |
|------------------------------------|---------------|---|---|
| (ATC level 1) | (ATC level 4) | N | % |

| | Total (N=XX) | |
|--------------------------|--------------|---|
| | N | % |
| Number of Systems (ATC1) | | |
| 1 | | |
| 2 | | |
| 3 | | |
| > 3 | | |
| Number of agents (ATC4) | | |
| 1 | | |
| 2 | | |
| 3 | | |
| > 3 | | |

Programming Notes: Percentage is based on total patient included.

Table 12.5.1. 3. Concomitant therapy during treatment. Summary of systems involved (ATC1).

| N | Median | Min | Max | Mean | SD* |
|---|---|---|---|---|---|
| (*) SD stands for standard devia | ation | | | | |
| Table 12.5.1. 4. Concomitant therapy | during treatment. Sur | mmary of agents i | involved (ATC4 | .). | |
| ${f N}$ | Median | Min | Max | Mean | SD |

| Table 12.5.1. 5. Listing of | Baseline characteristics: | Concomitant therapy. |
|---|---|---|
|---|---|---|

| Patient ID | Start date | ATC code | Route | •••• | Reason for use |
|------------|------------|----------|-------|------|----------------|

# 13 Figures.

**NOTE:** Figures will be showed for "all evaluable patients" and "all treated patients" by group when applicable. Also in case of patients with STR individual figures for the specific toxicity will be shown.

Figure 13. 1. Overall survival.



Figure 13. 2. Progression-free survival.







Kaplan-Meier curve of duration of response (If any response is observed).

Figure 13. 4. CA-125 for responders.



Figure 13. 5. Waterfall plots.



Maximum tumor shrinkage in measurable lesions by RECIST will be displayed. Additional graphs by tumour type and RECIST/CA-125 response will also be provided when applicable.

Figure 13. 6. Boxplot of LVEF evolution from BL .



Boxplot showing the change by cycle in LVEF from baseline.